CLINICAL TRIAL: NCT01918514
Title: The Effect of Adding Magnesium Sulfate to Standard Epidural and Interscalene Block in Treatment of Patients With Chronic Pain
Status: No longer available | Type: Expanded Access
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 455904-3
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2013-08

CONDITIONS: Pain
Keywords: Magnesium sulfate; epidural; interscalene; NMDA receptor
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: Adding Magnesium Sulfate to the standard epidural and interscalene blocks for chronic pain

SUMMARY:
Regional anesthesia is a safe, inexpensive technique, with the advantage of prolonged pain relief.

In the pain clinic the investigators perform different injections as the standard treatment for chronic pain based on the diagnosis and indications. Local anesthetic like Bupivacaine with or without Steroids (Depo-medrol) is used for these injections.

The investigators' goal is comparing pain control in different groups adding the magnesium sulfate 100mg to our compounds as an inexpensive, effective, and safe adjuvant to prolong the duration of analgesia and reduce the amount of narcotic dose.

DETAILED DESCRIPTION:
N-methyl-D-aspartate(NMDA) receptors are fundamental factors in controlling synaptic plasticity and memory function and play an important role in transition of acute pain to chronic intractable pain.

Magnesium is physiologic NMDA receptor antagonist. It will stabilized NMDA receptor and prevents influx of calcium and sodium ion. It has been studied that serum magnesium level is low in patients with chronic pain. Several studies has been done and shown that Magnesium has a significant effect in neuroprotection and membrane stabilization. Blocking the NMDA receptor will prevent activation of first order neurons in periphery or second order neurons in dorsal horn of spinal cord and then higher pain pathways to third order neurons and centers of the pain perception. Topical, oral and more effectively intravenous administration of magnesium has been used widely in treatment of chronic pain. There are limitations of intravenous administration of magnesium secondary to systemic cardiovascular side effects.

In several standardized study it has been shown that using magnesium intrathecally, epidurally or with interscalene injections can boost up the effect of opioids or local anesthetics. At the dose of 100 mg, it has been safe and effective to use.

Regional anesthesia is a safe, inexpensive technique, with the advantage of prolonged pain relief.

In the pain clinic the investigators perform different injections as the standard treatment for chronic pain based on the diagnosis and indications. Local anesthetic like Bupivacaine with or without Steroids (Depo-medrol) is used for these injections.

The investigators' goal is comparing pain control in different groups adding the magnesium sulfate 100mg to our compounds as an inexpensive, effective, and safe adjuvant to prolong the duration of analgesia and reduce the amount of narcotic dose. The investigators want to conduct a prospective, randomized, double-blind placebo controlled study with two major injections (2 different studies with the same concept):

1. Interscalene injection (2 subgroups including A: with Bupivacaine 0.25%(20ml) which is the standard injection with 1ml saline as placebo vs B: Bupivacaine 0.25%(20ml)+ Magnesium sulfate (100mg in 1 ml)
2. Epidural injection(2 subgroups including A:Bupivacaine 0.125%(8ml)+ Depo medrol(80mg) as the standard injection with 1ml saline as placebo vs B: Bupivacaine 0.125%(8ml)+ Depo medrol(80mg)+ Magnesium sulfate (100mg in 1 ml)

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 yrs of age and older
* Minimal level of pain of equal or higher than 4 out of 10 on Numerical Rating Scale(NRS=>4)
* The rest of inclusion criteria are based on pain clinic protocols for regular injections

Exclusion Criteria:

* Pregnant patients
* Children
* The rest of exclusion criteria are based on pain clinic protocols for regular injections

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: P. Sebastian Thomas, MD, Principal Investigator — SUNY Upstate UH
Locations (1):
- Upstate Comprehensive Pain Medicine Center, East Syracuse, New York, United States